CLINICAL TRIAL: NCT02140892
Title: A Comparison Study of Two Respiratory Physical Therapy Methods and Standard Medical Treatment for Treating COPD Patients During Acute Exacerbation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHEBA-13-0697-YO-CTIL
Record Dates: First submitted 2014-05-14; First posted 2014-05-16 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-05

CONDITIONS: Chronic Obstructive Pulmonary Disease; Chronic Bronchitis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- respiratory physical therapy manual technique (Experimental): respiratory physical therapy manual technique- Autogenic Drainage
  Interventions: Procedure: respiratory physical therapy manual technique- Autogenic Drainage
- respiratory physical therapy technique- IPV (Experimental): respiratory physical therapy technique- Intrapulmonary Percussive Ventilation
  Interventions: Device: respiratory physical therapy technique- IPV
- standart medical care (No Intervention): standard medical care

INTERVENTIONS:
Procedure: respiratory physical therapy manual technique- Autogenic Drainage
  Arms: respiratory physical therapy manual technique
Device: respiratory physical therapy technique- IPV
  Arms: respiratory physical therapy technique- IPV

SUMMARY:
One of the main goals of the respiratory physical therapy is to help people who are suffering from accumulating of secretions in their airways and lungs.

Chronic Obstructive Pulmonary Disease (COPD) patients are often hospitalized with an Acute Exacerbation of their medical condition.

Those patients usually get only the standard medical care during the acute phase and don't get respiratory physical therapy treatment.

The study's main aim is to investigate if respiratory physical therapy treatment in addition to standard medical care during the acute phase, can improve the respiratory and medical condition and reduce hospitalization stay.

In order to do so we will compare three groups of COPD patients during acute exacerbation; two groups will get one out of two respiratory physical therapy techniques; manually or Intrapulmonary Percussive Ventilator (IPV) in addition to standard medical care and the third group will get standard medical care alone.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of Acute Exacerbation of COPD or Acute Exacerbation of Chronic Bronchitis
* Respiratory Rate>25
* PaCO2> 45 mmHg
* 7.35 < PH < 7.38

Exclusion Criteria:

* intubation
* apnea
* glasgow coma scale < 8
* pneumothorax
* FEV1 < 50% predicted
* Ischemic Hearth Disease

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-07 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
length of stay in the hospital | up to three months